CLINICAL TRIAL: NCT04473573
Title: Spartan Cube CYP2C19 Inter Laboratory Reproducibility Study
Brief Title: Spartan Cube CYP2C19 Inter Laboratory Reproducibilty Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spartan Bioscience Inc. (Industry)
Collaborators: Children's Hospital of Eastern Ontario (Other); The Ottawa Hospital (Other); The University of Ottawa Heart Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: VNV-00227
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Genotyping Techniques
Keywords: Reproducibility of Results; CYP2C19

STUDY DESIGN:
Intervention Model Description: All subjects receive the same number and type of test for the duration of the study.
Who Masked: Participant, Investigator
Masking Description: Bi-directional sequencing results will not be shard with the participants, operators or Principal investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lot to Lot Reproducibility (Other): The purpose of this arm is to provide evidence to support that each lot of manufactured reagents for the Spartan Cube CYP2C19 Test produce the same result. Each participant, over the course of the study at the various sites, will be tested using 3 different lots of manufactured Spartan CYP2C19 Test Kits.
  Interventions: Device: Spartan Cube CYP2C19 System
- Site to Site Reproducibility (Other): The purpose of this arm was to provide supporting evidence that showed the same samples (subjects), when tested at different locations, produce the same result.
  Interventions: Device: Spartan Cube CYP2C19 System
- Operator Reproducibility (Other): The purpose of this arm was to provide supporting evidence that showed the same samples (subjects), when collected and tested by different operators, produce the same result.
  Interventions: Device: Spartan Cube CYP2C19 System

INTERVENTIONS:
Device: Spartan Cube CYP2C19 System — Using buccal material, determine the genotype of the *2, *3 and *17 SNPs of the CYP2C19 gene on the Spartan Cube CYP2C19 System.

SUMMARY:
The study verifies that the Spartan Cube CYP2C19 System generates reproducible results under multi-variant conditions including test site (three different test sites), operators (two operators per site), testing days (five non-consecutive days per site), and test kit lot (three different lots).

DETAILED DESCRIPTION:
The reproducibility study (VNV-00227) is aimed at assessing the performance of the Spartan Cube CYP2C19 product under multi-variant conditions that include test site, operators, testing days, and reagent lots. The sections below address how these variables were tested.

This study will be performed by a total of six operators at three test sites. At each site, two operators will conduct buccal sample collection and analysis. Operators include individuals who are technologists, technicians, and/or nurses. The buccal samples will be loaded in the Cube within one hour after buccal swab collection. Furthermore, results will be generated using multiple platforms (Spartan Cube, computer, and printer) and the same platforms will be used at each site. At each site, a total of 64 (8 subjects/operator x 2 operators x 2 sessions x 2 sub-sessions (replicates)) tests will be run on five non-consecutive days. Each day includes 2 sessions and 2 sub-sessions (total 4 collection times) in which samples will be collected. Test subject to platform pairing is not required, results will be generated on one of the platforms per session. This means that each site will generate a total of 320(64 obs./day x 5 days) results over the entire duration of the study.

To determine lot-to-lot reproducibility of test kits, three different lots will be evaluated. For this, two lots will be tested at each site. Each operator will use two lots per session on each testing day. Each replicate only includes a single lot of test kits.

All results generated by the Spartan Cube CYP2C19 System will be compared with the bi-directional sequencing results.

ELIGIBILITY:
Inclusion Criteria:

* available for travel to three different sites, on 5 non-consecutive days.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
% Agreement of test results generated on the Spartan Cube CYP2C19 System and bidirectional sequencing | Through study completion; anticipated to be less than 6 months
  Determine % agreement across all tests conducted and bi-directional sequencing results

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa Ahmed, PhD, Principal Investigator — Spartan Bioscience
Locations (3):
- Canada (3):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - The Univeristy of Ottawa Heart Institute, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No